CLINICAL TRIAL: NCT04643873
Title: Effects of Physical Activity Counseling and Pilates Exercises on Metabolic Control Variables in Patients With Prediabetes and Type 2 Diabetes:Randomised Controlled Study
Brief Title: Effects of Physical Activity in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, merve şuay üçgül, principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 13022260-300-95767
Record Dates: First submitted 2020-10-04; First posted 2020-11-25 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; PreDiabetes
Keywords: exercise; diabetus mellitus; type 2; counseling; prediabetic state
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): physical activity counseiling +pilates exercise group
  Interventions: Other: physical activity counseiling +pilates exercise group
- Experimental group 2 (Experimental): only physical activity counseiling group
  Interventions: Behavioral: physical activity counseiling group
- Control Group (No Intervention): only followed by family physician

INTERVENTIONS:
Other: physical activity counseiling +pilates exercise group — It is planned to do the pilates exercises for 50 minutes a day, 2 days a week during 12 weeks with physiotherapist. Pilates group patient will make pilates exercise once a week alone During physical activity counseling, considering the current physical and metabolic status of the person, the person-based 5A model of ACSM will be adapted to individuals with diabetes and physical activity consultancy will be provided
  Other Names: exercise
  Arms: Experimental group 1
Behavioral: physical activity counseiling group — During physical activity counseling, considering the current physical and metabolic status of the person, the person-based 5A model of ACSM will be adapted to individuals with diabetes and physical activity consultancy will be provided. Patients make aerobic and strengthening exercises by theirself based on phyiotherapist's suggestions
  Arms: Experimental group 2

SUMMARY:
The primary aim of our study is to evaluate the effects of physical activity counseling and pilates exercises on metabolic control variables in patients with prediabetes and type 2 diabetes; Its secondary aim is to examine the effects of both practices on physical activity level, exercise capacity and quality of life, and to compare the relationship between those under medical supervision by family doctor.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), diabetes is defined as a disease that occurs when the insulin hormone which is responsible for regulating blood glucose and secreted by the pancreas. It cannot be produced individually or used effectively by the body. It is a chronic disease with high morbidity and mortality and adversely affected by diabetes complications. Purpose in diabetes treatment; control of the individual's blood glucose level, prevention or control of complications. From the moment of diagnosis, healthy lifestyle changes are recommended for metabolic control in individuals with diabetes. Diabetes is classified as type 1, type 2, other specific causes and gestational diabetes according WHO. 90-95% of diabetes cases diagnosed all over the world are type 2 diabetes, 5-10% is type 1 diabetes and 2-3% is other diabetes types.

During exercise, oxygen and glucose input to muscle cells increases and regular physical activity provides metabolic control. Many studies have shown that physical activity has a protective effect on impaired glucose tolerance and prevents the risk of cardiovascular diseases and premature death in patients with type 2 diabetes. However, 60-70% of individuals with type 2 diabetes can not reach their daily physical activity goal and most of them can not maintain their regular exercise program. In order to prevent patients from giving up exercise early, it is important to provide personal counseling at certain periods, to encourage, support and advice during exercises, and to explain the exercises in a way that patients can understand.

In our study, patients with type 2 diabetes will be randomly divided into 3 groups as physical activity counseling and pilates exercise group, only physical activity counseling group, and control followed only with family physician recommendations and follow-up. It is planned to do the pilates exercises for 50 minutes a day, 2 days a week during 12 weeks with physiotherapist. Pilates group patient will make pilates exercise once a week alone. Individual exercise sessions will start with 5-10 minutes of warm-up exercises and end with cool-down exercises in the same time. Overall in the program; stretching exercises in different positions (standing and lying), exercises to increase the flexibility of the trunk muscles, upper extremity movements with and without an exercise ball, strengthening exercises with theraband will be applied. Types of movements to strengthen all abdominal muscles, muscles around the hips, back muscles, muscles in the shoulder girdle (shoulder bridge, corkscrew, roll-up, roll down, clam, side kick, staggered legs, scissors, swimming, swan dive, breast stroke preparation, Abdominal preparation, oblique preparation) will be used alternately in different sessions, from easy to difficult. Pilates exercises will be performed with light and relaxing music.

Within the scope of physical activity, moderate and / or high intensity aerobic exercise recommended by cIntegrating physical activity in primary care practice. The American Journal of Medicine (ACSM) will be recommended 150 minutes in a week. Care will be taken not to take a break for more than 2 days between two exercise days. In addition, strengthening exercises that will maintain or increase muscle strength including large muscle groups at least 3 days a week will be determined in accordance with the patient's current possibilities. Recommendations will be given for possible complications such as hypoglycemia during and after exercise.

During physical activity counseling, considering the current physical and metabolic status of the person, the person-based 5A model of ACSM will be adapted to individuals with diabetes and physical activity consultancy will be provided. The 5A model consists of assess, advise, agree, assist, and arrange subsections.

1. Assess: The person's level of knowledge about physical activity and diabetes, his perspective on exercise, his exercise history, readiness for change, fatigue, personal history and family history, and drug use will be evaluated. By asking open-ended questions, his attitude towards exercise will be determined.
2. Advise: The benefits of physical activity and the risks of physical inactivity will be explained, morbidities that may develop due to diabetes, the relationship of diabetes with physical activity, and exercise types will be mentioned. Short-term and long-term effects of exercise will be explained.
3. Agree: Cooperation will be made with the client in line with the person's wishes, interests and physical activity goals. Environmental resources for physical activity will be evaluated and appropriate guidance will be made. OMRON HJ 109 brand pedometer will be used for determining, monitoring and improving the level of physical activity.
4. Assist: Misunderstanding situations will be explained by helping the person identify and solve their problems with physical activity. Potential resources park, gym, etc., solutions will be produced together for the obstacles on the way to physical activity.
5. Arrange: A follow-up meeting will be held with the client one day a week, and the target will be determined for the next week. At the end of the interviews, the situation is summarized and it is aimed to increase clarity. During the interviews, motivational interview technique will be applied by the consultant, and a person-centered approach will be provided by establishing empathy.

Before and after the 12-week intervention program of all patients, metabolic control variables (body mass index, fasting blood glucose, HbA1c value, HDL, LDL, total cholesterol, triglyceride values) will be evaluated. Physical activity levels with IPAQ, exercise capacity with 6-minute walking test (6MWT), functional balance with Berg balance test and quality of life with SF-36 will be evaluated. Body fat percentage, visceral fat amount, body mass index and muscle mass amounts in the trunk and extremities will be calculated with the Jawon X-Contact 350 device. Exercise intensity during exercise will be determined by speaking test.

Metabolic control variables will be analyzed in the Healthy Life Park Blood Collection Unit affiliated to Iskenderun District Health Directorate after the permits are taken. Evaluation methods, exercise and consultancy applications will be carried out in Iskenderun Healthy Life Center. Only the participants in the family doctor follow-up will continue their routine doctor checks and recommendations.

An "Assessment Form" will be created to record the demographic and disease information of all cases included in the study. Diabetes year, prediabetes diagnosis time, history, family history, treatments taken, medications used, posture analysis with New York Posture Analysis, range of motion, muscle strength and shortness assessment and foot examination will be recorded in the evaluation form. Semmes Weinstein monofilament will be used for foot examination.

All analyzes will be performed using SPSS (Statistical Package for Social Sciences) for Windows 22. The compliance of the data to normal distribution will be evaluated by drawing the Kolmogorov-Smirnov test and histogram. Parametric tests will be used for data suitable for normal distribution. Data that are not suitable for normal distribution will be analyzed with non-parametric tests. Variables will be defined by their mean and standard deviation values. Analyzes and correlations between groups will be examined separately with appropriate tests. A value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with prediabetes or Type II diabetes at most 10 years ago
* Not using insulin
* Being under the age of 70
* Be woman
* Individuals regulated by glucose control, medication and / or diet
* Volunteering to exercise at least 3 days a week in the intervention group within the scope of the research
* Being able to communicate in Turkish written and verbal

Exclusion Criteria:

* Having uncontrolled hypertension (160/90 mmHg), cardiovascular problem, renal disease, neuropathy, systemic disease that will create contraindications for exercise
* Body mass index over 35 kg / m²
* Being a communication problem, not being able to cooperate

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
fasting blood glucose | up to 12 weeks
  A fasting blood sugar level less than 100 mg/dL (5.6 mmol/L) is normal. A fasting blood sugar level from 100 to 125 mg/dL (5.6 to 6.9 mmol/L) is considered prediabetes. If it's 126 mg/dL (7 mmol/L) or higher on two separate tests, you have diabetes percentage of body fat, amount of visceral fat, body mass index: amount of muscle mass in the trunk and extremities
HbA1c | up to 12 weeks
  A hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin. Normal: HbA1c below 5.7% Prediabetes: HbA1c between 5.7% and 6.4% Diabetes: HbA1c of 6.5% or higher
HDL | up to 12 weeks
  HDL (high-density lipoprotein cholesterol) cholesterol: High density lipoprotein cholesterol.60 mg/dL (1.6 mmol/L) or above is desirable
LDL | up to 12 weeks
  LDL (low-density lipoprotein cholesterol) Adult - < 130 mg/dL is normal value for LDL. Low-density lipoprotein is a type of lipoprotein that consists of cholesterol (LDL cholesterol, LDL-C) and similar substances with a small amount of protein
total cholesterol | up to 12 weeks
  Total cholesterol a measure of the total amount of cholesterol in your blood. It includes both low-density lipoprotein (LDL) cholesterol and high-density lipoprotein (HDL) cholesterol. Less than 200 mg/dL is normal
triglyceride values | up to 12 weeks
  Triglycerides are a type of fat (lipid) found in blood. Normal is less than 150 milligrams per deciliter (mg/dL), or less than 1.7 millimoles per liter (mmol/L)
percentage of body fat | up to 12 weeks
  Body fat percentage will be calculated with the Jawon X-Contact 350 device
Muscle mass amounts in the trunk and extremities | up to 12 weeks
  Muscle mass amounts in the trunk and extremities will be calculated with the Jawon X-Contact 350.Muscle mass includes the skeletal muscles, smooth muscles such as cardiac and digestive muscles and the water contained in these muscles
Step number | up to 12 weeks
  Average one week steps before and after intervention will be calculated with OMRON HJ 109 pedometer

SECONDARY OUTCOMES:
Short version of IPAQ (International Physical Activity Questionnaire) | up to 12 weeks
  Short version of IPAQ will be used to measure physical activity level
  . There are three levels of physical activity proposed to classify populations - 'low', 'moderate', and 'high' Vigorous Intensity = 8.0 METs Moderate Intensity = 4.0 METs
SF36 (Short Form 36) | up to 12 weeks
  SF36 will be used to measure quality of life Scoring between 0-100 High score means higher quality of life
6 minutes walk test | up to 12 weeks
  6 minutes walk test will be used to measure exercise capacity The six minute walk distance in healthy adults has been reported to range from 400m to 700m Age and sex-specific reference standards are available and may be helpful for interpreting 6MWT scores for both healthy adults and those with chronic diseases 47 . However, it is difficult to use normative values because of the differing methods used in studies. An improvement of 54m has been shown to be a clinically important difference24 in a study of people with chronic lung disease which is similar to the recommended criteria of meaningful clinical change of 50m based on analyses from a sample of 692 community living older adults and individuals who have survived a stroke 25
BMI (body mass index) | up to 12 weeks
  Weight and height will be combined to report BMI in kg/m^2. Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9. Obesity = BMI of 30 or greater
amount of visceral fat | up to 12 weeks
  Amount of visceral fat will be calculated with the Jawon X-Contact 350 device. Visceral fat is wrapped around major organs like the liver, pancreas and your kidney. Visceral fat ensures that there is some distance between each organ. Too much visceral fat creates can lead to inflammation and high blood pressure, which increases the risk of serious health problems. This is also know as central obesity.
  Based on all the available information Jawon X Contact 350 device gives you a range between 1 and 59. A rating between 1 and 12 indicates that you have a healthy level of visceral fat. A rating between 13 and 59 indicates that you have an excessive level of visceral fat.
Berg Balance Scale | up to 12 weeks
  The Berg Balance Scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait
waist circumference | up to 12 weeks
  Waist circumference is measured halfway between the lower ribs and the iliac crest
hip circumference | up to 12 weeks
  hip circumference is measured at the largest circumference around the buttocks
Waist-Hip Circumference Ratio | up to 12 weeks
  The waist-hip ratio is a simple technique for determining body fat distribution

CONTACTS AND LOCATIONS:
Overall Officials: ela tarakcı, prof dr, Study Chair — Istanbul University- Cerrahpasa Physiotherpy and Rehabilitation Department
Locations (1):
- Merve Suay, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Integrating Physical Activity in Primary Care Practice — https://pubmed.ncbi.nlm.nih.gov/26953063/
- See also: WHO Global report on diabetes: A summary. International Journal of Noncommunicable Diseases. 2016;1(1):3. — https://www.ijncd.org/article.asp?issn=2468-8827;year=2016;volume=1;issue=1;spage=3;epage=8;aulast=Roglic
- See also: Combined exercise for people with type 2 diabetes mellitus: a systematic review — http://pubmed.ncbi.nlm.nih.gov/22981711/